CLINICAL TRIAL: NCT02844998
Title: The Impact and Benefit of Physical Activity on Premature Ejaculation: Results of a Prospective, Randomized, Placebo-controlled Trial
Brief Title: The Impact and Benefit of Physical Activity on Premature Ejaculation
Acronym: PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, M.D., Ankara Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 5191
Record Dates: First submitted 2016-07-13; First posted 2016-07-26 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Premature Ejaculation
Keywords: intravaginal ejaculatory latency time; international physical activity questionnaire; premature ejaculation diagnostic tool
MeSH Terms: conditions — Premature Ejaculation | interventions — Exercise; dapoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dapoxetine 30 mg (Active Comparator): Patients who have sedentary life style will treat with Dapoxetine 30 mg (on demand)
  Interventions: Drug: dapoxetine 30 mg on demand
- Moderate Running (Experimental): Patients who have sedentary life style will be advised moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week. (Minimally active category)
  Interventions: Behavioral: physical activity
- Sham-controlled (Sham Comparator): Patients who have sedentary life style will be advised those to walk (not running )at most 30 minutes for 5 days in a week. (Inactive category)
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: physical activity — patients will do moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week
  Arms: Moderate Running; Sham-controlled
Drug: dapoxetine 30 mg on demand — Dapoxetine, a short-acting selective serotonin reuptake inhibitors, has been utilized for the treatment of premature ejaculation in various countries
  Arms: Dapoxetine 30 mg

SUMMARY:
The purpose of this study is to investigate the relationship between physical activity and PE, and determine whether moderate physical activity might delay ejaculation time or be an alternative treatment for PE.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active, heterosexual patients without regular physical activity or erectile dysfunction, and had a sexual partner for at least six months, and sexual intercourse at least twice a week

Exclusion Criteria:

* Use of medications for endocrinological, metabolic, chronic systemic, or psychiatric diseases, use of alcohol or addictive substances, or use of drugs that might affect erection and ejaculation, presence of patients with Peyronie's disease, chronic prostatitis, urethritis, or active urinary tract infection, and absence of regular physical activity or previous treatment for premature ejaculation.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Symonds T, Perelman MA, Althof S, Giuliano F, Martin M, May K, Abraham L, Crossland A, Morris M. Development and validation of a premature ejaculation diagnostic tool. Eur Urol. 2007 Aug;52(2):565-73. doi: 10.1016/j.eururo.2007.01.028. Epub 2007 Jan 16. PMID 17275165
- [Background] Sunay D, Sunay M, Aydogmus Y, Bagbanci S, Arslan H, Karabulut A, Emir L. Acupuncture versus paroxetine for the treatment of premature ejaculation: a randomized, placebo-controlled clinical trial. Eur Urol. 2011 May;59(5):765-71. doi: 10.1016/j.eururo.2011.01.019. Epub 2011 Jan 18. PMID 21256670

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Patients who have sedentary life style will treat with Dapoxetine 30 mg (on demand)
  dapoxetine 30 mg on demand: Dapoxetine, a short-acting selective serotonin reuptake inhibitors, has been utilized for the treatment of premature ejaculation in various countries
- Group 2: Patients who have sedentary life style will be advised moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week.
  Physical activity: patients will do moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week (To increase the physical activity level to "minimally active category or moderate physical activities [600-3,000 MET-min/week] according to IPAQ classification)
- Sham-controlled: Patients who have sedentary life style will be advised those to walk at most 30 minutes for 5 days in a week.
  physical activity: patients will do moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week. (inactive category [<600 MET-min/week] according to the IPAQ classification)
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Sham-controlled
Started | 42 | 39 | 39
Completed | 35 | 35 | 35
Not Completed | 7 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Patients who have sedentary life style will be advised moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week
  physical activity: patients will do moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week
- Sham-controlled: Patients who have sedentary life style will be advised those to walk at most 30 minutes for 5 days in a week.
  physical activity: patients will do moderate running which make them breathe somewhat harder than normal for at least 30 minutes for 5 days in a week
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Sham-controlled | Total
Number analyzed (Participants) | 35 | 35 | 35 | 105
Age, Categorical [Count of Participants; unit: Participants]
  Male: <=18 years | 0 | 0 | 0 | 0
  Male: Between 18 and 65 years | 35 | 35 | 35 | 105
  Male: >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35 | 35 | 35 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: count of participants] — All participitants are male
  count of participants
    Turkey | 35 | 35 | 35 | 105

OUTCOME MEASURES:

1. Primary Outcome: Premature Ejaculation Diagnostic Tool (Total Score)
Description: Premature Ejaculation Diagnostic Tool (PEDT) includes five items; control, frequency, minimal stimulation, distress, and interpersonal difficulty. In this classification tool, equal to or less than scores 8 indicates no PE, scores 9 and 10 indicate possible PE, and scores equal or higher than 11 indicates PE. Total score is between 2 and 22.
Time Frame: Baseline and 30 Days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 | Group 2 | Sham-controlled
Number analyzed (Participants) | 35 | 35 | 35
scores on a scale
  baseline data | 14.5 (1.9) | 13.7 (1.8) | 13.7 (2.2)
  end of study data | 8.9 (2.5) | 7.8 (2.9) | 12.8 (1.7)

2. Primary Outcome: Intravaginal Ejaculatory Latency Time
Description: Duration determined by the sexual partner with stopwatch method, and <1 minute was considered as PE. (minimum/maximum scores were not possible)
Time Frame: Baseline and 30 Days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group 1 | Group 2 | Sham-controlled
Number analyzed (Participants) | 35 | 35 | 35
seconds
  baseline data | 36.8 (13.1) | 39.3 (8.8) | 33.8 (14.7)
  end of study data | 181.7 (88.8) | 188.6 (82.9) | 50.3 (19.1)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Sham-controlled
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No